CLINICAL TRIAL: NCT00190320
Title: Induction of Labor or Waiting for Suspicion Fetal Macrosomia (DAME)
Brief Title: DAME: Induction of Labor or Waiting for Suspicion Fetal Macrosomia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe AUCAN, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P030417
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2007-03

CONDITIONS: Fetal Macrosomia
Keywords: Fetal macrosomia; Neonatal traumatism; Maternal morbidity
MeSH Terms: conditions — Fetal Macrosomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Induction of labor vs waiting

SUMMARY:
Aim of the study :The major aim is to evaluate the effectiveness of the induction of labor in case of fetal macrosomia on the reduction of neonatal traumatism risk. The secondary aims are to evaluate maternal morbidity and the risk of Caesarean in case of induction of labor, compared to a spontaneous labor.

DETAILED DESCRIPTION:
A clinical trial multicentric randomized controlled will be organized. A total of 1000 women will be recruited between 36 and 38 weeks of amenorrhoea (GW) if the pregnancy is single, in cephalic presentation and the fetus is estimated macrosomic for the gestational age (> 90e percentile clinically and >95° percentile sonographically).All agreeing patients will be randomized in one of the two following groups: - 1. Induction of labor between 37+0 and 38+6 GW and within 3 day after the randomization. - 2. Expectancy until the spontaneous beginning of labor or up to 41 GW.The measurement of principal exit is the neonatal traumatism (criterion composite associating: dystocia of the shoulders, fractures osseous, paralysis/paresis of the plexus brachial or intracerebral haemorrhage).The secondary criteria are neonatal asphyxiation (arterial pH < 7.10 or Apgar < 7 to 5 minutes), the maternal traumatism (tear of 3rd or 4th degree) and the Caesarean. The long-term after-effects for the mother and her child will be also evaluated

ELIGIBILITY:
Inclusion Criteria:

* Agreed women Sonographic estimation of begin of pregnancy <20GW Single pregnancy in cephalic presentation Macrosomic fetus :
* clinical estimation : 36GW : ≥3350g or 34cm 37GW : ≥3550gor34cm 38GW : ≥3750g or 35cm
* sonographic estimation : 36GW : ≥ 3500g 37GW : ≥ 3700g 38GW : ≥ 3900g

Exclusion Criteria:

* Typical diabetes I or typifies II or diabetes gestational treated by insulin.
* Antecedents of tear of the anal sphincter or severe urinary or faecal presence of an incontinence.
* Antecedent of dystocia of the shoulders or neonatal traumatism.
* Antecedents of caesarian or uterine scar.
* contraindication in the release of the work or in the childbirth by low way.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2005-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
reduction of neonatal traumatism risk | 52 months

SECONDARY OUTCOMES:
reduction of maternal morbidity and caesarean | 52 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick ROZENBERG, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHI Poissy st Germain, Poissy, France

REFERENCES:
- [Derived] Boulvain M, Thornton JG. Induction of labour at or near term for suspected fetal macrosomia. Cochrane Database Syst Rev. 2023 Mar 8;3(3):CD000938. doi: 10.1002/14651858.CD000938.pub3. PMID 36884238
- [Derived] Boulvain M, Senat MV, Perrotin F, Winer N, Beucher G, Subtil D, Bretelle F, Azria E, Hejaiej D, Vendittelli F, Capelle M, Langer B, Matis R, Connan L, Gillard P, Kirkpatrick C, Ceysens G, Faron G, Irion O, Rozenberg P; Groupe de Recherche en Obstetrique et Gynecologie (GROG). Induction of labour versus expectant management for large-for-date fetuses: a randomised controlled trial. Lancet. 2015 Jun 27;385(9987):2600-5. doi: 10.1016/S0140-6736(14)61904-8. Epub 2015 Apr 8. PMID 25863654